CLINICAL TRIAL: NCT03415763
Title: Efficacy of Adjuvant Chemotherapy in Patients With Clinical Stage III Rectal Cancer Undergoing Neoadjuvant Chemoradiotherapy: A Pathology-oriented, Prospective, Multicenter, Randomized, Open-label, Parallel Group Clinical Trial
Brief Title: Adjuvant Chemotherapy in Patients With Clinical Stage III Rectal Cancer Undergoing Neoadjuvant Chemoradiotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: LI XIN-XIANG (Other)
Responsible Party: Sponsor-Investigator, LI XIN-XIANG, Professor, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fudan AC
Record Dates: First submitted 2018-01-17; First posted 2018-01-30 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Rectal Neoplasms
Keywords: Rectal Neoplasms; Adjuvant Chemotherapy; Neoadjuvant Chemoradiotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Observation (No Intervention): Observation for patients with pathological complete response or yp stage I(According to the postoperative pathological stage, the present study was designed as a non-inferiority trail for patients with pathological complete response or yp stage I to compare the long-term outcomes of observational group and those receiving 5-fluorouracil)
- 5-fluorouracil (Experimental): Capecitabine for patients with pathological complete response or yp stage I Capecitabine 1250 mg/m2 twice daily for 14 days in a 3-week cycle to be administered orally after food, three cycles(According to the postoperative pathological stage, the present study was designed as a non-inferiority trail for patients with pathological complete response or yp stage I to compare the long-term outcomes of observational group and those receiving 5-fluorouracil )
  Interventions: Drug: Capecitabine
- 5-fluorouracil alone (Experimental): 5-fluorouracil alone for patients with yp stage II or III Capecitabine 1250 mg/m2 twice daily for 14 days in a 3-week cycle to be administered orally after food, three cycles(According to the postoperative pathological stage, the present study was designed as a superiority trail for patients with yp stage II or III to compare the effect of oxaliplatin combined with 5-fluorouracil and 5-fluorouracil alone)
  Interventions: Drug: Capecitabine
- mFOLFOX6 or CAPOX (Experimental): Oxaliplatin combined with 5-fluorouracil for patients with yp stage II or III mFOLFOX6 (leucovorin 400 mg/m2 as a 2-hour infusion, and the concurrent administration of oxaliplatin 85 mg/m2 as a 2-hour infusion, followed by a bolus of 5-FU 400 mg/m2 within 15 min and 46-hour infusion of 5-FU 2400 mg/m2 on day 1 every 2 weeks), three cycles or CAPOX (oxaliplatin 130 mg/m2 as a 2-hour infusion on day 1, followed by capecitabine 1000 mg/m2 twice daily for 14 days every 3 weeks), three cycles( According to the postoperative pathological stage, the present study was designed as a superiority trail for patients with yp stage II or III to compare the effect of oxaliplatin combined with 5-fluorouracil and 5-fluorouracil alone)
  Interventions: Drug: mFOLFOX6 or CAPOX

INTERVENTIONS:
Drug: Capecitabine — According to the postoperative pathological stage, the present study was designed as a non-inferiority trail for patients with pathological complete response or yp stage I to compare the long-term outcomes of observational group and those receiving 5-fluorouracil. For patients with yp stage II or III, the study aims to compare the effect of oxaliplatin combined with 5-fluorouracil and 5-fluorouracil alone.
  Other Names: Xeloda
  Arms: 5-fluorouracil; 5-fluorouracil alone
Drug: mFOLFOX6 or CAPOX — According to the postoperative pathological stage, the present study was designed as a non-inferiority trail for patients with pathological complete response or yp stage I to compare the long-term outcomes of observational group and those receiving 5-fluorouracil. For patients with yp stage II or III, the study aims to compare the effect of oxaliplatin combined with 5-fluorouracil and 5-fluorouracil alone.
  Other Names: 5-Fu-leucovorin-oxaliplatin or xeloda-oxaliplatin
  Arms: mFOLFOX6 or CAPOX

SUMMARY:
The purpose of this study is to evaluate the efficacy of adjuvant chemotherapy in patients with clinical stage III rectal cancer who received neoadjuvant chemoradiotherapy on the basis of postoperative pathological stage.

DETAILED DESCRIPTION:
Previous studies have proved that neoadjuvant radiotherapy can decrease the rate of local recurrence rather than distal metastases in advanced rectal cancer. Moreover, the local control was not responsible for survival benefit. Adjuvant chemotherapy is capable of eliminating the micrometastasis, rendering better prognosis to rectal cancer. However, the application of adjuvant chemotherapy depends largely on the evidence from colon cancer. At present, controversy remains on the clinical value of adjuvant chemotherapy in patients with rectal cancer who received neoadjuvant chemoradiotherapy. Besides that, the pathological stage followed by neoadjuvant chemoradiotherapy may have an effect on the evaluation of adjuvant chemotherapy. According to the postoperative pathological stage, the present study was designed as a non-inferiority trail for patients with pathological complete response or yp stage I to compare the long-term outcomes of observational group and those receiving 5-fluorouracil. For patients with yp stage II or III, the study aims to compare the effect of oxaliplatin combined with 5-fluorouracil and 5-fluorouracil alone.

ELIGIBILITY:
Inclusion Criteria:

* The lesion must be within 12 cm of the anus as measured by endoscopy
* Histologically confirmed diagnosis of rectal carcinoma
* CT, MRI and EUS verified as clinical stage III rectal cancer without involvement of other organs
* Without multiple primary cancer
* Sufficient organ function
* Able to provide written informed consent

Exclusion Criteria:

* Younger than 18 years or older than 75 years
* Synchronous or metachronous malignancy within 5 years.
* Patients with Intestinal obstruction or perforation or bleeding who require emergency surgery.
* Patients with a history of pelvic irradiation.
* ASA grade IV or V.
* Women who are pregnant (confirmed by serum b-HCG in women of reproductive age) or breast feeding.
* Severe mental illness.
* Patients with severe emphysema, interstitial pneumonia, or ischemic heart disease who can not tolerate surgery.
* Patients who received steroid therapy within one month.
* Patients or family members misunderstand the conditions and goals of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 764 (Estimated)
Dates: Start 2018-11-05 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 3-year
  Calculated from the date of surgery to the date of recurrence

SECONDARY OUTCOMES:
Overall survival | 3-year, 5-year
  Calculated from the date of diagnosis to the date of death from any cause
Disease free survival | 5-year
  Calculated from the date of surgery to the date of recurrence
The rate of local recurrence | 3-year
  The ratio of the number of local recurrence to the total patients
The rate of adverse events resulted from chemotherapy | 3-year
  The ratio of the number of patients experienced adverse events to the total patients
The quality of life postoperatively | 3-month, 6-month, 9-month, 12-month, 18-month, 24-month
  The European Organization for Research and Treatment (EORTC)-QLQ-C30 HRQL questionnaire was assessed with repeated measures at regular intervals postoperatively at months 3, 6, 9, 12, 18, and 24

CONTACTS AND LOCATIONS:
Overall Officials: Xinxiang Li, MD,PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li Q, Luo D, Zhu J, Yang L, Liu Q, Ma Y, Liang L, Cai S, Zhang Z, Li X; ACRNaCT study group. ACRNaCT trial protocol: efficacy of adjuvant chemotherapy in patients with clinical T3b/T4, N+ rectal Cancer undergoing Neoadjuvant Chemoradiotherapy: a pathology-oriented, prospective, multicenter, randomized, open-label, parallel group clinical trial. BMC Cancer. 2019 Nov 15;19(1):1117. doi: 10.1186/s12885-019-6289-6. PMID 31729964